CLINICAL TRIAL: NCT00844415
Title: Open-label Safety and Tolerability Study of Dabigatran Etexilate Mesilate Given for 3 Days at the End of Standard Anticoagulant Therapy in Children Aged 12 Years to Less Than 18 Years
Brief Title: Safety and Tolerability of Dabigatran Etexilate in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160.88
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2013-03-26 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran

ARMS (1):
- dabigatran etexilate (Experimental): open label; patient to receive dabigatran etexilate BID for three days
  Interventions: Drug: dabigatran etexilate

INTERVENTIONS:
Drug: dabigatran etexilate — 2.14 mg/kg BID to a max 150 mg BID

SUMMARY:
To investigate the safety and tolerability of dabigatran etexilate capsules in a small group of eight adolescent patients.

ELIGIBILITY:
Inclusion criteria:

1. males or females 12 to less than 18 years of age
2. objective diagnosis of primary VTE
3. completion of planned treatment course with LMWH or OAC for primary VTE
4. written informed consent by parent (legal guardian) and patient assent

Exclusion criteria:

1. weight less than 32 kg
2. conditions associated with increased risk of bleeding
3. severe renal dysfunction or requirement for dialysis
4. active infective endocarditis
5. hepatic disease
6. pregnant females or females not using medically accepted contraceptive method
7. anemia or thrombocytopenia
8. use of prohibited or restricted drug within previous week
9. received investigational drug within past 30 days
10. unreliable patients or patients who have any condition that would not allow safe participation in study

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2012-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Canada (2):
  - 1160.88.00002 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1160.88.00001 Boehringer Ingelheim Investigational Site, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Halton JM, Lehr T, Cronin L, Lobmeyer MT, Haertter S, Belletrutti M, Mitchell LG. Safety, tolerability and clinical pharmacology of dabigatran etexilate in adolescents. An open-label phase IIa study. Thromb Haemost. 2016 Aug 30;116(3):461-71. doi: 10.1160/TH15-04-0275. Epub 2016 Jun 30. PMID 27357738

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients (Pat.): Dabigatran was administered twice daily for three consecutive days (total 6 doses). All patients received an initial oral dose of 1.71mg/kg of dabigatran (80 percent of the adult dose of 150 mg/70 kg adjusted for the patient's weight). Based on thrombin time (TT) and clinical assessment, the dose was adjusted to the target dose of 2.14 mg/kg of dabigatran (100 percent of the adult dose adjusted for the patient's weight). Three patients received 75 mg dabigatran (first dose) followed by 100 mg twice daily (BID). Three patients took dabigatran 100 mg (first dose) followed by 125 mg BID. Two patients received a dose of 125 mg dabigatran followed by 150 mg BID. One patient received only a single dose of dabigatran (75 mg).
Period: Overall Study
Arm/Group | All Patients (Pat.)
Started | 9 (Entered and treated.)
Pat. Received 75mg Followed by 100mg | 3
Pat. Received 100mg Followed by 125mg | 3
Pat. Received 125mg Followed by 150mg | 2
Pat. Received Single Dose 75mg | 1
Completed | 8 (Completed.)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- All Patients: Dabigatran was administered twice daily for three consecutive days (total 6 doses). All patients received an initial oral dose of 1.71mg/kg of dabigatran (80 percent of the adult dose of 150 mg/70 kg adjusted for the patient's weight). Based on thrombin time (TT) and clinical assessment, the dose was adjusted to the target dose of 2.14 mg/kg of dabigatran (100 percent of the adult dose adjusted for the patient's weight). Three patients received 75 mg dabigatran (first dose) followed by 100 mg twice daily (BID). Three patients took dabigatran 100 mg (first dose) followed by 125 mg BID. Two patients received a dose of 125 mg dabigatran followed by 150 mg BID. One patient received only a single dose of dabigatran (75 mg).
Arm/Group | All Patients
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Bleeding Events (Major and Minor)
Description: Patients were carefully assessed for signs and symptoms of bleeding. Bleeding was to be classified as major or minor. Major bleeding had to satisfy one or more of the following criteria:
  Overt bleeding associated with a decrease in haemoglobin of at least 2 g/dL in 24 hours, Overt bleeding requiring a transfusion of red blood cells, Overt bleeding which was retroperitoneal, intracranial, intraocular, or intraarticular, any overt bleeding deemed by the attending physician to require discontinuation of study medication. Minor bleeds were clinical bleeds that did not fulfill the criteria for major bleeds.
Time Frame: From Screening until 30 days after first drug administration (end of trial visit)
Population: Treated set (TS). This patient set includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Measure: Number; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 9
Participants | 0

2. Primary Outcome: Number of Patients With Adverse Events
Description: Patients with treatment drug related adverse events (DRAEs) and serious adverse events (SAEs) are reported separately for on-treatment and post-treatment period. Events were considered "on-treatment" if occurring within 72 hours after last drug administration.
Time Frame: From Screening until 30 days after first drug administration (end of trial visit)
Population: TS
Measure: Number; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 9
Participants
  DRAEs on-treatment | 2
  SAEs on-treatment | 0
  DRAEs post-treatment | 0
  SAEs post-treatment | 1

3. Primary Outcome: Plasma Concentration of Free Dabigatran
Description: Plasma concentration of free dabigatran measured at 72 hours after first dose
Time Frame: 3 days
Population: Treated Set. Descriptive statistics for the concentration measurement could only be calculated for the subgroups of patients receiving the same sequence of doses. Statistics were only reported for groups with at least 3 patients (non-sparse data).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- All Patients: Dabigatran was administered twice daily for three consecutive days (total 6 doses). All patients received an initial oral dose of 1.71mg/kg of dabigatran (80 percent of the adult dose of 150 mg/70 kg adjusted for the patient's weight). Based on thrombin time (TT) and clinical assessment, the dose was adjusted to the target dose of 2.14 mg/kg of dabigatran (100 percent of the adult dose adjusted for the patient's weight). Three patients received 75 mg dabigatran (first dose) followed by 100 mg twice daily (BID). Three patients took dabigatran 100 mg (first dose) followed by 125 mg BID. However, for the two patients who received a dose of 125 mg dabigatran followed by 150 mg BID, and the one patient who received only a single dose of dabigatran (75 mg), no summary statistics were calculated, due to sparse data.
Arm/Group | All Patients
Number analyzed (Participants) | 6
ng/ml
  Patients with 75mg dose followed by 100mg (N=3) | 28.0 (12.8)
  Patients with 100mg dose followed by 125mg (N=3) | 41.6 (66.5)

4. Primary Outcome: Plasma Concentration of Total Dabigatran
Description: Plasma concentration of total dabigatran measured at 72 hours after first dose
Time Frame: Day 3
Population: TS with non-sparse data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | All Patients
Number analyzed (Participants) | 6
ng/ml
  Patients with 75mg dose followed by 100mg (N=3) | 34.2 (3.56)
  Patients with 100mg dose followed by 125mg (N=3) | 58.2 (48.7)

5. Primary Outcome: Thrombin Time (TT) Centrally Measured
Description: Measurement of TT was performed locally and centrally by Hemoclot Thrombin Inhibitor clotting assay.
Time Frame: Day 3
Population: TS with non-sparse data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | All Patients
Number analyzed (Participants) | 6
seconds
  Patients with 75mg dose followed by 100mg (N=3) | 36.9 (3.61)
  Patients with 100mg dose followed by 125mg (N=3) | 37.4 (3.97)

6. Primary Outcome: TT Locally Measured
Description: Measurement of TT was performed locally and centrally by Hemoclot Thrombin Inhibitor clotting assay.
Time Frame: Day 3
Population: TS with non-sparse data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | All Patients
Number analyzed (Participants) | 6
seconds
  Patients with 75mg dose followed by 100mg (N=3) | 33.5 (2.15)
  Patients with 100mg dose followed by 125mg (N=3) | 36.8 (5.72)

7. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT) Centrally Measured
Description: Measurement of aPTT was performed locally and centrally using validated assays.
Time Frame: Day 3
Population: TS with non-sparse data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | All Patients
Number analyzed (Participants) | 6
seconds
  Patients with 75mg dose followed by 100mg (N=3) | 38.6 (2.94)
  Patients with 100mg dose followed by 125mg (N=3) | 47.4 (4.42)

8. Secondary Outcome: aPTT Locally Measured
Description: Measurement of aPTT was performed locally and centrally using validated assays.
Time Frame: Day 3
Population: TS with non-sparse data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | All Patients
Number analyzed (Participants) | 6
seconds
  Patients with 75mg dose followed by 100mg (N=3) | 29.9 (2.68)
  Patients with 100mg dose followed by 125mg (N=3) | 33.6 (0.896)

9. Secondary Outcome: Ecarin Clotting Time (ECT)
Description: Measurement of ECT was performed locally and centrally using validated assays. Descriptive statistics is only performed for the centrally measured ECT.
Time Frame: Day 3
Population: TS with non-sparse data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | All Patients
Number analyzed (Participants) | 6
seconds
  Patients with 75mg dose followed by 100mg (N=3) | 43.3 (1.31)
  Patients with 100mg dose followed by 125mg (N=3) | 49.6 (11.6)

10. Secondary Outcome: Patients With Clinically Relevant Changes in Any Laboratory Parameter, Electrocardiogram (ECG) or Vital Signs
Description: Changes in any laboratory parameter, ECG or vital signs were judged clinically relevant by the investigator.
Time Frame: Baseline and 3 days
Population: TS
Measure: Number; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 9
Participants | 0

11. Secondary Outcome: Occurences of Clinical Outcome
Description: Occurrences of clinical outcomes including recurrent venous thrombolic event (VTE), post thrombotic syndrome (PTS), pulmonary emboli (PEs), and total and VTE related mortality objectively assessed for example by ultrasound, venography or computed chromatography (CT) scan (based on the thrombus location). Number of patients with particular clinical outcome are reported.
Time Frame: 3 days
Population: TS
Measure: Number; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 9
Participants
  Patients with recurrent VTE | 1
  Patients with PTS | 0
  Patients with PE | 0
  Patients with VTE related death | 0
  Patients with other death | 0
  Patients with other clinical outcome | 0

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=9)
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.